CLINICAL TRIAL: NCT04698356
Title: Pilot Study - Validation of Speech Materials for an Auditory-cognitive Training Paradigm (NIH P01 Project - Speech Perception With High Cognitive Demand)
Brief Title: Speech Perception With High Cognitive Demand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Joe Smith, Director - HRPP (L. Decruy is no longer at UMD), University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P01AG055365 (NIH); P01AG055365 (NIH)
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Speech Intelligibility; Aging
Keywords: Auditory-cognitive training; Aging; Speech-in-noise perception
MeSH Terms: conditions — Speech Intelligibility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Validation of auditory-cognitive training paradigm (Experimental): In order to provide maximal speech-in-noise training benefit for older, normal-hearing adults, a validation of our new training materials is required. The investigators will evaluate the translated and adjusted sentences (based on the Nottingham UK PLUS training paradigm), the adaptive procedure, and the short-term memory component, in young, normal-hearing adults (18-30 years). Based on the results of this pilot study, the investigators can further optimize the sentences and procedures to be used during the training paradigm for older adults.
  Interventions: Behavioral: Auditory-cognitive training paradigm

INTERVENTIONS:
Behavioral: Auditory-cognitive training paradigm — The investigators developed an American English version of the Nottingham (UK) PLUS training paradigm in which listeners are asked to focus and listen to one speaker while ignoring another speaker. The paradigm is designed to optimally enhance the possibility of benefit: an adaptive procedure is employed in order to train each individual at their own level and to make the task challenging. A short-term memory component was also added to the original training paradigm, to enhance the cognitive skills of our participants. To provide maximal speech-in-noise benefit for older, normal-hearing adults, a validation of our new training materials is required. The investigators will evaluate this in young, normal-hearing adults (18-30 years) by studying our outcome measure (speech reception threshold) for the different sentence-scenarios and test-retest sessions.

SUMMARY:
With advancing age, adults experience increasing speech understanding difficulties in challenging situations. Currently, speech-in-noise difficulties are rehabilitated by providing hearing aids. For older normal-hearing adults, however, hearing devices do not provide much benefit since these adults do not have a decreased hearing sensitivity. The goal of the "Speech Perception with High Cognitive Demand" Project is to evaluate the benefit of a new auditory-cognitive training paradigm. In order to provide maximal benefit for older, normal-hearing adults, a validation of the new training materials is required. In a pilot study, the investigators will evaluate the new auditory-cognitive training paradigm in 15 young, normal-hearing adults (18-30 years). Based on these results, the training paradigm can be further optimized for older adults.

DETAILED DESCRIPTION:
With advancing age, adults experience increasing speech understanding difficulties in challenging situations, such as difficulty with understanding other persons in a noisy restaurant. Speech-in-noise difficulties are typically rehabilitated by providing hearing aids. For older normal-hearing adults, however, hearing devices do not provide much benefit since these adults do not have a decreased hearing sensitivity. For these adults communication difficulties persist in everyday life situations and can even lead to social withdrawal, isolation, and depression.

A growing body of studies demonstrates that combined auditory-cognitive training paradigms can offer speech-in-noise benefits to adults with hearing loss that could prevent the consequences listed above (Ferguson & Henshaw, 2015; Lawrence et al., 2018). The goal of the "Speech Perception with High Cognitive Demand" Project is to evaluate the benefit of a new auditory-cognitive training paradigm for older normal-hearing adults. The investigators developed an American English version of the Nottingham (UK) PLUS training paradigm in which listeners are asked to focus and listen to one speaker while ignoring another speaker. Although it cannot ensured that every participant will experience direct significant benefit from the training, the paradigm is being designed to optimally enhance the possibility of benefit: an adaptive procedure is employed in order to train each individual at their own level and to make the task challenging, and a short-term memory component is added to the original training paradigm to also enhance the cognitive skills of the participants. In addition, the training is implemented on tablets rather than computers, making at-home training possible (many older adults are more comfortable with tablets than laptops). This way, not only the risk of COVID-19 for participants is minimized, but training is also provided in a realistic setting which will ensure a better transfer of the trained skills to daily communication situations.

In order to provide maximal benefit for older, normal-hearing adults, a validation of the new training materials is however required, and the initial validation will be for younger adults only. The investigators will evaluate the translated and adjusted sentences (from UK to American English), the adaptive procedure, and the short-term memory component, in young, normal-hearing adults (18-30 years). Based on the results of this pilot study, the sentences and procedures of the training paradigm can be further optimized for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-30 years
* Normal hearing (pure-tone thresholds <= 25 dB HL from 250-8000 Hz)
* Dominant language: American English
* Education: a high school diploma or higher educational level

Exclusion Criteria:

* Middle-ear or inner ear pathology
* Non-native speaker of English
* Inability to complete all training sessions within a pre-specified time window (e.g., due to unexpected schedule restrictions)
* Learning disorders.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Speech reception threshold (SRT) | Through study completion, an average of 2 months
  Sentences of seven different scenarios will be presented to young, normal-hearing adults. Participants will be instructed to listen to one speaker and ignore the other one, will be asked to recall the keywords of the to-be-attended sentence after the target sentence (0-back) or after the next sentence was presented (1-back; short-term memory component). The sentences will be presented using an 2 down-1up adaptive procedure in which the ratio of the levels of the to-be-attended and to-be-ignored speaker will be adjusted based on the correctly recalled keywords. This means that the procedure will converge to a level-ratio for which the participant understands 71% of the to-be-attended speaker, also called the speech reception threshold (SRT). The SRT will be used to compare the 0-back versus 1-back task and the validity of the different scenarios/sentences and procedures (mean/median SRT, inter- and intrasubject variability of the scenarios and test-retest session).

CONTACTS AND LOCATIONS:
Overall Officials: Samira B Anderson, PhD, Principal Investigator — University of Maryland, College Park; Jonathan Z Simon, PhD, Principal Investigator — University of Maryland, College Park; Stefanie E Kuchinsky, PhD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Department of Hearing and Speech Sciences, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Promotheus